CLINICAL TRIAL: NCT07271004
Title: Proprioceptive Training Reduces Headache Burden and Center of Pressure Path Length in Patients With Cervicogenic Headache: A Randomized Controlled Trial
Brief Title: Proprioceptive Training Reduces Headache Burden and Center of Pressure Path Length in Patients With Cervicogenic Headache
Acronym: PTRHBCOP-CGH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hungarian University of Sports Science (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelaziz Emam, Principal Investigator, Hungarian University of Sports Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003409
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache;; Headache Burden; Postural Balance; Proprioception; Eye Movements
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Proprioception

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated into two parallel groups with equal allocation (1:1 ratio). The control group received a standard physiotherapy program including heat therapy, TENS, ultrasound, and cervical mobility and strengthening exercises. The experimental group received the same physiotherapy program plus a 10-minute proprioceptive gaze direction recognition (GDR) training task during each session. Both groups underwent three sessions per week for eight weeks. The design allowed for comparison of outcomes between groups receiving standard therapy alone versus those receiving standard therapy combined with proprioceptive training.
Who Masked: Outcomes Assessor
Masking Description: Type: Single (Outcomes Assessor)
  Roles Masked: Outcomes Assessor
  Participant Masked: No
  Care Provider Masked: No
  Investigator Masked: No
  Outcomes Assessor Masked: Yes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive (Experimental): Participants in the experimental group received the same standard physiotherapy program as the control group, with the addition of a 10-minute proprioceptive Gaze Direction Recognition (GDR) training task during each session.
  The GDR training involved observing another person's head and neck rotations from behind and identifying the direction of gaze, requiring motor imagery and visuospatial judgment to activate cervical sensorimotor pathways. Task difficulty was progressively increased across sessions.
  Training was administered three times per week for eight weeks, each session lasting approximately 60 minutes.
  Interventions: Other: Proprioception
- Control Group (Active Comparator): Participants in the control group received a standardized physiotherapy program three times per week for eight weeks. Each 60-minute session included:
  20 minutes of moist heat applied to the neck and shoulder region,
  20 minutes of transcutaneous electrical nerve stimulation (TENS) at 50 Hz and 100 µs pulse width,
  5 minutes of continuous-mode ultrasound therapy (1-1.5 W/cm²) to the cervical muscles, and
  A series of therapeutic exercises to improve cervical mobility, posture correction, and neck-muscle strength through isometric contractions.
  This program represented the conventional physiotherapy regimen for cervicogenic headache management.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Proprioception — The GDR training involved observing another person's head and neck rotations from behind and identifying the direction of gaze, requiring motor imagery and visuospatial judgment to activate cervical sensorimotor pathways. Task difficulty was progressively increased across sessions.
  Training was administered three times per week for eight weeks, each session lasting approximately 60 minutes.
  Would you like me to now write the Intervention Description sections (the short entries that go under "Intervention Name," "Type," and "Description" linked to each arm)? Those are the next fields after the Arm descriptions.
  Arms: Proprioceptive
Other: Conventional physical therapy — 20 minutes of moist heat applied to the neck and shoulder region,
  20 minutes of transcutaneous electrical nerve stimulation (TENS) at 50 Hz and 100 µs pulse width,
  5 minutes of continuous-mode ultrasound therapy (1-1.5 W/cm²) to the cervical muscles, and
  A series of therapeutic exercises to improve cervical mobility, posture correction, and neck-muscle strength through isometric contractions.
  Arms: Control Group

SUMMARY:
Cervicogenic headache (CGH) is a secondary headache originating from dysfunction in the cervical spine and is associated with impaired sensorimotor control and postural instability. This randomized, assessor-blinded, parallel-group clinical trial aims to investigate whether adding gaze direction recognition (GDR)-based proprioceptive training to a conventional physiotherapy program can reduce headache burden and improve postural balance in individuals with CGH. Participants are randomly allocated to receive either standard physiotherapy or standard physiotherapy plus GDR training for eight weeks. Primary outcomes include headache frequency, headache duration, and center-of-pressure (COP) path length during quiet standing. The study is conducted in accordance with ethical guidelines and was approved by the relevant institutional review board.

DETAILED DESCRIPTION:
Cervicogenic headache (CGH) is a secondary headache arising from disorders of the cervical spine and related structures. Individuals with CGH commonly present with impaired cervical proprioception and altered postural control. Sensorimotor retraining strategies, such as gaze direction recognition (GDR), have been used in chronic neck pain populations to target proprioceptive deficits; however, their application in CGH has not been comprehensively investigated.

This randomized, controlled, assessor-blinded clinical trial is designed to evaluate whether adding proprioceptive GDR training to a standardized physiotherapy program results in greater reductions in headache burden and improvements in postural balance compared with physiotherapy alone. Thirty-eight participants meeting ICHD-3 diagnostic criteria for CGH are randomly assigned in a 1:1 ratio to a control group receiving standard physiotherapy or to a treatment group receiving standard physiotherapy plus GDR training. The intervention is delivered three times per week for eight weeks.

The standardized physiotherapy program includes thermotherapy, transcutaneous electrical nerve stimulation (TENS), ultrasound therapy, and therapeutic exercises for cervical mobility, posture correction, and isometric strengthening. The treatment group receives the same program with the addition of a structured GDR proprioceptive task.

Gaze Direction Recognition Exercise (GDRE) Procedure:

During the GDRE, the therapist sits in a chair positioned 0.75 m behind the center of a wooden table (1.8 × 0.4 × 0.76 m). Six wooden blocks, numbered 1 to 6 from left to right, are placed along the table edge nearest the therapist, spaced 0.31 m apart. Patients sit in a chair behind the therapist with a clear view of the numbered blocks.

An assistant signals the start of each trial, at which point the therapist randomly directs his gaze and head toward one of the blocks. As patients observe the therapist's neck rotation from behind, they rotate their own head in the same direction and verbally report the number of the block they believe the therapist is looking at. Patients are instructed to avoid moving other body parts during head rotation. No accuracy feedback is provided to the patient. The assistant records both reaction time and accuracy for each response. Each GDRE session consists of 30 trials and lasts approximately 10 minutes.

Primary outcomes include headache frequency (attacks per month), headache duration (hours per attack), and center-of-pressure (COP) path length during quiet standing, measured at baseline and after eight weeks of intervention. The study protocol was reviewed and approved by the Faculty of Physical Therapy Ethics Committee, Cairo University, and all participants provide written informed consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed cervicogenic headache (CGH) according to current diagnostic criteria
* Age 35 to 49 years
* Unilateral pain originating in the neck and radiating to the frontotemporal region
* Pain aggravated by neck movements
* Restricted cervical range of motion
* Joint tenderness in at least one upper cervical joint (C1-C3)
* Headache frequency of at least one episode per month for the past year

Exclusion Criteria:

* History of head or neck injury or surgery
* Musculoskeletal disorders
* Neurological diseases or disorders
* Metabolic syndromes
* Hypertension or hypotension
* Vestibular disorders
* Inner ear inflammation

Ages: 35 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Headache frequency (attacks per month) | Baseline and after 8 weeks of intervention
  Change in the number of cervicogenic headache attacks per month, as recorded by participants in a headache diary. Headache frequency was averaged over four weeks at baseline and again at post-intervention. Lower values indicate improvement.
Headache duration (hours per attack) | Baseline and after 8 weeks of intervention
  Change in the mean duration of headache episodes, expressed in hours per attack, recorded from participant headache diaries. Duration was averaged across all episodes within each 4-week period at baseline and post-treatment.

SECONDARY OUTCOMES:
Center of Pressure (COP) path length (cm) | Baseline and after 8 weeks of intervention
  Change in total center-of-pressure path length measured during quiet standing using the HUMAC Balance System (CSMi, USA). Shorter path length reflects improved postural stability and sensorimotor control.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy kfs university, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this study will be made available upon reasonable request. The shared dataset will include variables related to baseline demographics, group allocation, headache frequency, headache duration, and center-of-pressure (COP) path length outcomes. Data will be provided in a coded format without any information that could identify individual participants. Access will be granted to qualified researchers for academic and non-commercial purposes following approval of a methodologically sound proposal and signing of a data access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the main results and remain accessible for 3 years thereafter.
Access Criteria: Qualified researchers may request access to the de-identified dataset for the purpose of academic, non-commercial research related to cervicogenic headache, physiotherapy, or sensorimotor training. Requests should include a brief study proposal outlining objectives, methods, and data requirements. Access will be granted following review and approval by the principal investigator and after execution of a data access agreement ensuring participant confidentiality and compliance with ethical data use standards.

REFERENCES:
- [Background] Nobusako S, Matsuo A, Morioka S. Effectiveness of the gaze direction recognition task for chronic neck pain and cervical range of motion: a randomized controlled pilot study. Rehabil Res Pract. 2012;2012:570387. doi: 10.1155/2012/570387. Epub 2012 May 7. PMID 22645685